CLINICAL TRIAL: NCT03710122
Title: A Prospective, Randomized, Multi-centered, Placebo-controlled Clinical Trial of Oral Vanycomycin in Adults With Primary Sclerosing Cholangitis
Brief Title: Vancomycin for Primary Sclerosing Cholangitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Elizabeth Carey (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Carey, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-003439; FD-R-6102 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vancomycin (Experimental)
  Interventions: Drug: Vancomycin
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vancomycin — Firvanq by Azurity Pharmaceuticals, Inc.
  Arms: Vancomycin
Other: Placebo — Placebo for Vancomycin
  Arms: Placebo

SUMMARY:
To find out if vancomycin is a safe and effective therapy for primary sclerosing cholangitis.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
A. Determine if OV normalizes serum ALP in adults with PSC. Levels of serum ALP obtained at 6,12,and 18 months of OV treatment, and at 3, and 6 months post OV treatment will be compared to those obtained at baseline (month 0), and with values at the same study time points in the placebo arm.

B. Determine if OV stabilizes or improves liver fibrosis assessed by LSM using TE. Liver stiffness will be measured at 6, 12, and 18 months of OV treatment, and at 6 months post OV treatment, and values will be compared to those obtained at baseline (month 0), and with values in the placebo arm.

C. Determine the changes in the intestinal microbiota in relation to the use of OV, and study the correlation between the changes in the intestinal microbiota and the changes in: 1) liver enzymes, particularly serum ALP, and 2) liver stiffness, assessed by LSM using TE.

D. Determine if changes in proinflammatory cytokines (TGF-β, IL-4, IL-13, IL-10, etc.) predict response to OV. Cytokines will be measured at baseline, months 6, 12, 18, and at 3, and 6 months post OV treatment, if the study is positive.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject age 18-76 years
2. Diagnosis of PSC consistent with the guidelines published by the American Association for the Study of Liver Diseases (AASLD).39 All subjects must have an elevated serum ALP of at least 1.5 times upper limit of normal at baseline plus cholangiographic evidence of PSC, as demonstrated by magnetic resonance imaging, endoscopic retrograde cholangiography, direct cholangiography, or liver biopsy.
3. Total bilirubin at screening must be ≤ 2 times upper limit of normal
4. An ultrasound (or equivalent imaging modality) that excludes biliary obstruction and malignancy within 6 months of study entry,
5. If a patient is on any of the following medications and/or supplements, he or she is expected to remain on the same daily dose through the treatment period: UDCA, azathioprine, prednisone (or an equivalent steroid compound), methotrexate, a 5-aminosalicylic acid, biologic therapy, and/or a probiotic.
6. If a patient has been on obeticholic acid or other experimental therapies for PSC, they must complete a 3 month washout period before study entry
7. PSC with or without inflammatory bowel disease, such as ulcerative colitis or Crohn's disease
8. Must agree to comply with the study protocol and provide informed consent.

Exclusion Criteria:

1. Administration of an antibiotic within 3 months prior to the study,
2. Pregnancy or attempting to become pregnant or breastfeeding,
3. Presence of any of the following:

   i. Hepatitis B infection

   ii. Hepatitis C infection (antibody positive); patients with a history of hepatitis C infection will be eligible for this study if they have undetectable levels of HCV RNA

   iii. Other cholestatic liver diseases such as primary biliary cholangitis and cholestatic diseases of pregnancy

   iv. Metabolic liver diseases such as Wilson's disease and hemochromatosis

   v. Inherited diseases of the liver such as α-1 antitrypsin deficiency

   vi. Immunoglobulin G4-related cholangitis

   vii. PSC with concomitant autoimmune hepatitis (AIH) and/or primary biliary cholangitis (previously known as primary biliary cirrhosis)

   viii. Secondary sclerosing cholangitis (SSC),

   ix. Active acute ascending cholangitis requiring antibiotics

   x. CCA (malignant biliary stricture, neoplasm, and cytology/histopathology or positive fluorescence in situ hybridization (FISH) consistent with adenocarcinoma of the bile duct)

   xi. A liver biopsy, if one has been previously obtained, which showed non-alcoholic steatohepatitis (NASH). Patients with suspected fatty liver by imaging will not be excluded

   xii. Presence of decompensated cirrhosis such as hepatic encephalopathy, hepato-renal syndrome and hepato-pulmonary syndrome,

   xiii. History of liver transplantation, anticipated need for liver transplantation within 12 months from randomization, or a Model of End Stage Liver Disease (MELD) score of ≥15

   xiv. Ongoing alcohol abuse (>4 drinks per day for men, and >2 drinks per day for women)

   xv. History of allergic reaction to vancomycin,

   xvi. Moderate-to-severe renal impairment with a calculated creatinine clearance of < 60mL/min

   xvii. HIV/AIDS,

   xviii. Any other conditions or abnormalities that, in the opinion of the investigator, may compromise the safety of the subject or interfere with the subject participating in or completing the study.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Alkaline phosphatase at 6 months | 6 months
  Determine if OV normalizes serum ALP in adults with PSC. Levels of serum ALP obtained at 6 months of OV treatment, and will be compared to those obtained at baseline (month 0), and with values at the same study time points in the placebo arm.
Alkaline phosphatase at 12 months | 12 months
  Determine if OV normalizes serum ALP in adults with PSC. Levels of serum ALP obtained at 12 months of OV treatment, and will be compared to those obtained at baseline (month 0), and with values at the same study time points in the placebo arm.
Alkaline phosphatase at 18 months | 18 months
  Determine if OV normalizes serum ALP in adults with PSC. Levels of serum ALP obtained at 18 months of OV treatment, and will be compared to those obtained at baseline (month 0), and with values at the same study time points in the placebo arm.
Alkaline phosphatase at 3 months post treatment = 21 months | 21 months
  Determine if OV normalizes serum ALP in adults with PSC. Levels of serum ALP obtained at 3 months post OV treatment, and will be compared to those obtained at baseline (month 0), and with values at the same study time points in the placebo arm.
Alkaline phosphatase at 6 months post treatment = 24 months | 24 months
  Determine if OV normalizes serum ALP in adults with PSC. Levels of serum ALP obtained at 6 months post OV treatment, and will be compared to those obtained at baseline (month 0), and with values at the same study time points in the placebo arm.

SECONDARY OUTCOMES:
Fibroscan, cholangiography | 18 months
  Transient elastography (TE), a new technique that allows non-invasive assessment and follow up of liver fibrosis by measuring liver stiffness, differentiates between severe from non-severe fibrosis in PSC, and the rate of progression of liver stiffness measurement (LSM) assessed by TE correlates well with the rate of progression of fibrosis in PSC and with patients' clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Carey, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Arizona State University, Tempe, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials